CLINICAL TRIAL: NCT02572245
Title: A Phase 1, Open-label, Randomized, Single Dose, Parallel Group Comparability Study To Assess The Pharmacokinetics Of Pf-06410293 Following Subcutaneous Administration Using A Prefilled Syringe Or A Prefilled Pen In Healthy Adult Subjects
Brief Title: A Study of PF-06410293 Following Subcutaneous Administration Using A Prefilled Syringe Or A Prefilled Pen In Healthy Adult Subjects
Acronym: B538-05
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: B5381005
Record Dates: First submitted 2015-09-25; First posted 2015-10-08 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-06

CONDITIONS: Healthy Subjects
Keywords: Healthy Subjects; Device; PK; Phase 1; Bioequivalence; Adalimumab; Single Dose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-06410293 PFS (Prefilled Syringe) (Active Comparator): PF-06410293 40 mg administered by Prefilled Syringe (PFS)
  Interventions: Device: PF-06410293 PFS
- PF-06410293 PFP (Prefilled Pen) (Active Comparator): PF-06410293 40 mg administered by Prefilled pen
  Interventions: Device: PF-06410293 PFP

INTERVENTIONS:
Device: PF-06410293 PFS — PF-06410293 40 mg administered subcutaneously by Prefilled syringe
  Arms: PF-06410293 PFS (Prefilled Syringe)
Device: PF-06410293 PFP — PF-06410293 40 mg administered subcutaneously by prefilled pen
  Arms: PF-06410293 PFP (Prefilled Pen)

SUMMARY:
This is a study comparing adalimumab Pfizer (PF-06410293) administered as a subcutaneous(SC) injection using a pre-filled syringe (PFS) or pre-filled pen in healthy adult subjects

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female subjects and/or male subjects, who, at the time of screening, are between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, complete physical examination including blood pressure and pulse rate measurement, 12 lead electrocardiogram (ECG), and clinical laboratory tests.
2. Body Mass Index (BMI) of 17.5 to 32 kg/m2; and a total body weight >50 kg (110 pounds).
3. Chest X ray with no evidence of current, active TB or previous (inactive) TB, fungal or general infections, heart failure, malignancy, or other clinically significant abnormalities taken at Screening or within 24 weeks prior to Day 1 and read by a qualified radiologist.
4. Female subjects of non childbearing potential must meet at least one of the following criteria: a. Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; status may be confirmed by having a serum follicle stimulating hormone (FSH) level confirming the post menopausal state; b. Have undergone a documented hysterectomy and/or bilateral oophorectomy; c. Have medically confirmed ovarian failure.

All other female subjects (including females with tubal ligations) will be considered to be of childbearing potential.

Exclusion Criteria:

1. Evidence or history of clinically significant infectious, hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, autoimmune, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
2. Evidence or history of nervous system demyelinating diseases (including multiple sclerosis, optic neuritis, Guillain Barré syndrome).
3. History of relevant orthostatic hypotension, fainting spells or blackouts.
4. Previous history of cancer, except for adequately treated basal cell or squamous cell carcinoma of the skin

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 164 (Actual)
Dates: Start 2016-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Maximum serum concentration (Cmax) | Day 1 - Day 15
Area under the concentration curve (AUC 0-2wk) | Day 1-Day 15

SECONDARY OUTCOMES:
Injection site tolerability (Subject Assessment - Visual Analog Scale) - Mean Injection site pain over 24 hour period post dose | Hour 0 (immediately after injection), 15 minutes, 1, 3, 8, 12 and 24 hours post injection
  Mean injection site pain over a 24 hour period post dose rated by subject on a visual analog scale (VAS), compared for injection by PFS or PFP, and for the 2 injection locations using each device
Injection site tolerability (Blinded Safety Assessor - Modified Draize Scale) - Mean injection site tolerability over 24 hour post dose | 1, 3, 8, 12 and 24 hours post injection
  Mean injection site tolerability using the Modified Draize Scale Numerical Grade over 24 hours post dose rated by the blinded Safety Assessor, compared for injection by PFS or PFP, and for the 2 injection locations using each device
Time to reach the maximum serum concentration (Tmax) | Day 1 - Day 43
AUC from time 0 to the last time point with quantifiable concentration (AUCT) | Day 1 - Day 43
AUC extrapolated to infinity (AUC0 inf) | Day 1 - Day 43
Volume of distribution (Vz/F), | Day 1 - Day 43
Apparent clearance (CL/F) | Day 1 - Day 43
Terminal half life (t1/2) | Day 1 - Day 43

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- ICON Early Phase Services, LLC, San Antonio, Texas, United States

REFERENCES:
- [Derived] Cox DS, Alvarez DF, Bock AE, Cronenberger CL. Randomized, Open-Label, Single-Dose, Parallel-Group Pharmacokinetic Study of PF-06410293 (adalimumab-afzb), an Adalimumab Biosimilar, by Subcutaneous Dosing Using a Prefilled Syringe or a Prefilled Pen in Healthy Subjects. Clin Pharmacol Drug Dev. 2021 Oct;10(10):1166-1173. doi: 10.1002/cpdd.939. Epub 2021 Mar 25. PMID 33765358
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5381005&StudyName=A%20Phase%201%2C%20Open-label%2C%20Randomized%2C%20Single%20Dose%2C%20Parallel%20Group%20Comparability%20Study%20To%20Assess%20The%20Pharmacokinetics%20Of%20Pf-06410293%20Following%20Subcutaneous%20Administration%20Using%20A%20Prefilled%20Syringe%20Or%20A%20Prefilled%20Pen%20In%20Healthy%20Adult%20Subjects
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5381005&StudyName=A+Phase+1%2C+Open-label%2C+Randomized%2C+Single+Dose%2C+Parallel+Group+Comparability+Study+To+Assess+The+Pharmacokinetics+Of+Pf-06410293+Following+Subcutaneous+Administration+Using+A+Prefilled+Syringe+Or+A+Prefilled+Pen+In+Healthy+Adult+Subjects